CLINICAL TRIAL: NCT04954053
Title: Validity and Reliability of the Turkish Version of Wheelchair User's Shoulder Pain Index
Brief Title: The Turkish Version of the WUSPI
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Şeyda ÖZAL, Research Assistant, Gazi University
Other Study IDs: Gazi Uni
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Shoulder Pain
Keywords: Wheelchair User; WUSPI; Turkish version; Validity and Reliability
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Wheelchair users frequently experience shoulder pain. It has been determined that in our country, the subjective assessment methods that will help to determine and monitor shoulder pain severity of wheelchair users are limited. The purpose of this study is to adapt the original English version of the Wheelchair Users Shoulder Pain Index into Turkish and to assess its validity and reliability.

Firstly, the original English version of WUSPI was translated into Turkish and culturally adapted, then applied to 100 wheelchair users to investigate the validity of the scale. The reliability of the scale was assessed by internal consistency and test-retest analysis and found a high internal consistency. Validation of WUSPI-Tr was assessed by the concurrent validity method. To establish concurrent validity, WUSPI scores were compared to SPADI and ASES scores by Spearman correlation analysis. There was a positively excellent correlation with SPADI and, negatively excellent correlation with ASES. As a result, it is determined tath the Turkish version of WUSPI-Tr is a valid and reliable tool.

DETAILED DESCRIPTION:
The original version of WUSPI was translated into Turkish via multistep translation rules. It is culturally adapted into Turkish. The semantic equivalence of the new scale was evaluated and the Turkish version of the WUSPI (WUSPI-Tr) has been created. It is applied to 100 wheelchair users to investigate the validity of the scale. People who are at least for 1 year using a manual wheelchair as their primary means of mobility, cognitively unimpaired, literate, and older than 18 years are included in this study. The reliability of the scale was assessed by internal consistency and test-retest analysis. As a result of the analysis, the Cronbach Alfa value was calculated as 0.894, and WUSPI-Tr was found to have high internal consistency. The WUSPI-Tr questionnaire was re-administered to 50 participants for 7 to 14 days for the test-retest method and the results were compared with the Interclass Correlation Coefficient (ICC) method. WUSPI has been found to have high reliability (0.997). Validation of WUSPI-Tr was assessed by the concurrent validity method. To establish concurrent validity, WUSPI scores were compared to SPADI and ASES scores by Spearman correlation analysis. The correlation coefficient of WUSPI-Tr with SPADI is 0.931 and with ASES was -0.812. These results show that there was a positively excellent correlation with SPADI and, negatively excellent correlation with ASES (p < 0,001). As a result, the Turkish version of WUSPI-Tr is a valid and reliable tool.

ELIGIBILITY:
Inclusion Criteria:

* accepting the participation
* using manual wheelchairs as the primary mobility tool for more than a year

Exclusion Criteria:

* being illiterate,
* having cognitive impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult wheelchair users who used manual wheelchairs as the primary mobility tool for more than a year
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-02-05 (Actual); Primary Completion 2017-04-26 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Wheelchair User's Shoulder Pain Index | First Day
  self-reported outcome measure
Shoulder Pain and Disability Index (SPADI) | First Day
  self-reported outcome measure
The Society of American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES) | First Day
  self-reported outcome measure
Wheelchair User's Shoulder Pain Index | 2 weeks later
  self-reported outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Şeyda ÖZAL, MSc, Principal Investigator — Gazi University Faculty of Health Sciences Physiotherapy and Rehabilitation Department; Selda Başar, Assoc Prof, Study Director — Gazi University Faculty of Health Sciences Physiotherapy and Rehabilitation Department; Nevin Ergun, Prof Dr, Study Chair — Sanko University Faculty of Health Sciences Physiotherapy and Rehabilitation Department
Locations (1):
- Gazi University Faculty of Health Sciences Physioteraphy and Rehabilitation Department, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the corresponding author upon reasonable request.

REFERENCES:
- [Background] Gellman H, Sie I, Waters RL. Late complications of the weight-bearing upper extremity in the paraplegic patient. Clin Orthop Relat Res. 1988 Aug;(233):132-5. PMID 3402118
- [Background] Curtis KA, Black K. Shoulder pain in female wheelchair basketball players. J Orthop Sports Phys Ther. 1999 Apr;29(4):225-31. doi: 10.2519/jospt.1999.29.4.225. PMID 10322595
- [Background] Finley MA, Rodgers MM. Prevalence and identification of shoulder pathology in athletic and nonathletic wheelchair users with shoulder pain: A pilot study. J Rehabil Res Dev. 2004 May;41(3B):395-402. doi: 10.1682/jrrd.2003.02.0022. PMID 15543457
- [Background] Curtis KA, Roach KE, Applegate EB, Amar T, Benbow CS, Genecco TD, Gualano J. Development of the Wheelchair User's Shoulder Pain Index (WUSPI). Paraplegia. 1995 May;33(5):290-3. doi: 10.1038/sc.1995.65. PMID 7630657
- [Background] Curtis KA, Roach KE, Applegate EB, Amar T, Benbow CS, Genecco TD, Gualano J. Reliability and validity of the Wheelchair User's Shoulder Pain Index (WUSPI). Paraplegia. 1995 Oct;33(10):595-601. doi: 10.1038/sc.1995.126. PMID 8848314
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Snyder CF, Aaronson NK, Choucair AK, Elliott TE, Greenhalgh J, Halyard MY, Hess R, Miller DM, Reeve BB, Santana M. Implementing patient-reported outcomes assessment in clinical practice: a review of the options and considerations. Qual Life Res. 2012 Oct;21(8):1305-14. doi: 10.1007/s11136-011-0054-x. Epub 2011 Nov 3. PMID 22048932
- [Background] Weir JP. Quantifying test-retest reliability using the intraclass correlation coefficient and the SEM. J Strength Cond Res. 2005 Feb;19(1):231-40. doi: 10.1519/15184.1. PMID 15705040